CLINICAL TRIAL: NCT05641766
Title: Multimodal Magnetoencephalography and Electroencephalography Exploration of the Acute Effects of THC Exposure on Neural Noise and Information Transmission Within Working Memory Networks
Acronym: THC-MEG
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Jose Cortes, Assistant Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2000033383; 1R03DA054453-01A1 (NIH)
Record Dates: First submitted 2022-11-29; First posted 2022-12-08 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: THC
Keywords: MEG; EEG; THC; Placebo; Working Memory; Neural Noise; Cognitive Process
MeSH Terms: interventions — Dronabinol

STUDY DESIGN:
Intervention Model Description: This proof-of-concept study will use a double-blind, randomized, cross-over (within-subject), placebo-controlled, counterbalanced study design in which participants will receive 0 (placebo) or 0.03 mg/kg intravenous THC over 20 minutes while undergoing simultaneous MEG/EEG data collection.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- THC (Experimental): Participants will receive THC into a rapidly flowing IV infusion.
  Interventions: Drug: THC
- Placebo (Other): Participants will receive an equivalent amount (about 1-2 ml) of placebo (sterile 190 proof USP ethanol). The placebo does not produce any measurable blood alcohol levels or subjective/behavioral effects.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: THC — Participants will receive THC into a rapidly flowing IV infusion.
  Arms: THC
Other: Placebo — Participants will receive an equivalent amount (about 1-2 ml) of placebo (sterile 190 proof USP ethanol). The placebo does not produce any measurable blood alcohol levels or subjective/behavioral effects.
  Arms: Placebo

SUMMARY:
The purpose of this study is to use non-invasive brain imaging methods (MEG and EEG) to characterize the effects of THC on brain activity during learning.

DETAILED DESCRIPTION:
The goal of this study is to use multimodal MEG/EEG to gain novel insight into the acute effects of THC on neural noise and its interaction with the fast information processing dynamics of the brain's cognition-related functional neural networks.

ELIGIBILITY:
Inclusion Criteria:

* Cannabis use at least once in the past 12 months
* No cannabis use during the course of the study confirmed with negative urine toxicology at screening and on each test day
* Good physical and mental health

Exclusion Criteria:

* Cannabis naïve individuals
* Lifetime or current medical, psychiatric or psychosocial disorders or history that is deemed unsuitable for participation in the study per PI discretion.
* Positive pregnancy test, lactation, or refusal to practice birth control for the duration of the study and for two weeks following completion
* Major current or recent stressors
* Positive urine drug test
* Contraindication for Magnetic Resonance Imaging
* Treatment with psychotropic medication as per discretion of the PI
* IQ less than 80
* Weight exceeding 166kg
* Diagnosis of major psychotic or manic disorder in first-degree relatives.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-31 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Changes in brain dynamics during the Sternberg Working Memory Task | Baseline and starting at +15 minutes after start of IV THC or placebo administration
  Changes in brain dynamics will be characterized during the Sternberg Working Memory Task where participants are presented with a list of items to memorize, followed by a memory maintenance period during which the subject must maintain the list of items in memory.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | Baseline and starting at +15 minutes after start of IV THC or placebo administration
  To confirm the acute effects of THC, feeling states associated with cannabis intoxication will be measured using a self-reported visual analogue scale of four feeling states ("high","anxious","calm and relaxed", and "tired") associated with cannabis effects. Subjects will be asked to score the perceived intensity of these feeling states at that moment on a 11mm line from 0=not at all to 100=extremely.
Clinician Administered Dissociative Symptoms Scale (CADSS) | Baseline and starting at +15 minutes after start of IV THC or placebo administration
  To confirm the acute effects of cannabis, perceptual alterations will be measured using the CADSS. This is a scale consisting of 19 self-report items and 8 clinician-rated items scored 0=not at all to 4=extremely. The scale captures alterations in environmental/time/body perception, feelings of unreality, and memory impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Cortes-Briones, PhD, Principal Investigator — Yale University
Locations (1):
- VA Connecticut Healthcare System, Yale School of Medicine, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No